CLINICAL TRIAL: NCT07345377
Title: Exploratory Clinical Study to Investigate the Therapeutic Mechanisms, Efficacy Prediction, and Safety Profile of Individualized Transcranial Magnetic Stimulation as a Therapeutic Intervention in Adult Participants Diagnosed With Irritable Bowel Syndrome, Utilizing Multimodal Magnetic Resonance Imaging for Neuroimaging Assessment and High-Throughput Sequencing for Fecal Microbiota Analysis and Metabolic Profile Detection
Brief Title: Study on Treatment Mechanisms and Efficacy Prediction of Individualized Transcranial Magnetic Stimulation in Adults With Irritable Bowel Syndrome Using Multimodal MRI and High-Throughput Sequencing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024(E2)-HS-009
Record Dates: First submitted 2025-12-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Irritable Bowel Syndrome (IBS); Pain; Depressive Disorder, Major, Moderate
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain; Depressive Disorder; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This study adopts a parallel group design, with participants randomly assigned to either the individualized TMS intervention group or the sham-TMS control group. The two groups are compared simultaneously to evaluate the efficacy and safety of the intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized TMS Intervention (Experimental): Participants in this group receive the individualized transcranial magnetic stimulation (TMS) intervention.
  Interventions: Device: Individualized TMS Intervention
- Sham TMS Intervention (Sham Comparator): Participants in this group receive the sham TMS intervention (for blinding purposes).
  Interventions: Device: Sham TMS Intervention

INTERVENTIONS:
Device: Individualized TMS Intervention — This individualized transcranial magnetic stimulation (TMS) intervention distinguishes itself from conventional fixed-target TMS by using resting-state fMRI functional connectivity to determine the personalized left dorsolateral prefrontal cortex (DLPFC) target. It uses a Magstim TMS system (infrared optical navigation) for precise positioning. Stimulation intensity is 90% of the individual's resting motor threshold (RMT; MEPs >50μV in ≥5/10 stimulations), delivered via the iTBS paradigm (3 pulses/burst [50Hz], 5Hz burst repetition, 2s stimulation/8s rest, 3 cycles/1800 pulses per session). This personalized targeting design enhances precision, setting it apart from non-individualized TMS in other studies.
  Arms: Individualized TMS Intervention
Device: Sham TMS Intervention — This sham TMS intervention is designed to maintain double-blinding: it uses the same equipment (Magstim infrared navigation TMS system), procedures (individual RMT measurement, personalized left DLPFC target positioning), iTBS paradigm (3 pulses/burst [50Hz], 5Hz repetition, 2s/8s cycle, 1800 pulses/session) and duration (20min core/40min total per session, 10 total sessions) as the individualized TMS in this study. Its only distinction (from the experimental intervention) is the 90° coil orientation (directing magnetic field away from the scalp, no effective cortical stimulation).
  Arms: Sham TMS Intervention

SUMMARY:
The goal of this clinical trial is to explore if "individualized repetitive Transcranial Magnetic Stimulation (TMS)" works to improve symptoms in adults with Irritable Bowel Syndrome (IBS). It also aims to learn how this treatment works (by looking at links between the brain, gut, and gut bacteria) and if tests like brain scans or gut bacteria checks can show if the treatment will work for a person. The main questions it aims to answer are:

Will individualized TMS improve IBS symptoms (like stomach pain or discomfort) and affect the links between the brain, gut, and gut bacteria? Can brain scan results (from multimodal Magnetic Resonance Imaging, MRI) and gut bacteria checks (from high-throughput sequencing) predict how well a person responds to TMS?

Participants will be adults aged 18-59 who:

Meet the Rome Ⅳ criteria for IBS (a standard way to diagnose IBS); Have stopped taking IBS-related medicines for more than 2 weeks; Do NOT have MRI or TMS contraindications (like metal implants in the body, mental illness, pregnancy, or serious illnesses requiring hospital stays).

Participants will:

Receive 10 TMS sessions (5 times a week, for 2 weeks total) - TMS is a non-invasive treatment that uses gentle magnetic pulses on the scalp;

Before the first TMS session, and again after the 10th session:

Fill out surveys to rate IBS symptoms; Have an MRI scan (painless, takes about 60 minutes) to look at brain activity; Provide a small stool sample to check gut bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Rome IV diagnostic criteria for Irritable Bowel Syndrome (IBS);
* Has discontinued IBS-related medications for more than 2 weeks prior to enrollment;
* Aged between 18 and 75 years (inclusive);
* Has sufficient cognitive ability to provide informed consent, understand study instructions, and complete questionnaires.

Exclusion Criteria:

* Has contraindications to MRI (e.g., metal implants in the body, claustrophobia) or TMS (e.g., history of epilepsy, skull defects);
* Diagnosed with mental illnesses (e.g., schizophrenia, bipolar disorder) that require ongoing medication or psychotherapy;
* Women who are pregnant, breastfeeding, or planning to become pregnant during the study period;
* Presents signs of severe illness requiring hospitalization (e.g., hemodynamic instability, acute infection, acute myocardial infarction, cerebral infarction);
* Has taken any substances that may affect study indicators (e.g., probiotics, prebiotics) within 3 months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Rating Scale (IBS-SSS) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assessment of the severity of irritable bowel syndrome symptoms (including abdominal pain, bloating, diarrhea/constipation, and impact on daily life) using the IBS-SSS. Scale Details: Minimum value: 0 points; Maximum value: 500 points; Score interpretation: Higher scores indicate more severe IBS symptoms.
17 items-Hamilton Depression Rating Scale (HAMD-17) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assessment of the severity of depressive symptoms in participants using the 17-item Hamilton Depression Rating Scale. Scale Details: Minimum value: 0 points; Maximum value: 54 points; Score interpretation: Higher scores indicate more severe depressive symptoms.
14 items-Hamilton Anxiety Rating Scale (HAMA-14) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assesses the severity of anxiety symptoms in participants, covering both psychological anxiety dimensions (e.g., tension, fear, restlessness) and somatic anxiety dimensions (e.g., palpitations, muscle soreness, gastrointestinal discomfort). Scale Details: Minimum value: 0 points; Maximum value: 56 points; Score interpretation: Higher scores indicate more severe anxiety symptoms.
Brain Structure Features (Multimodal MRI) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assessment of brain structural indicators including gray matter volume (measured by voxel-based morphometry) and white matter integrity (measured by fractional anisotropy via diffusion tensor imaging).
Brain Function Features (Multimodal MRI) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assessment of brain functional indicators covering multiple dimensions of neural activity and circuit organization:
  * Spontaneous brain activity: Quantifies the intensity and synchronization of intrinsic resting-state neural activity, including: Amplitude of low-frequency fluctuations (ALFF); Regional Homogeneity (ReHo).
  * Functional connectivity: Measures inter-regional neural associations, including: Seed-based correlation analysis; Dynamic Causal Modeling (DCM).
  * Brain network organization: Analyzes large-scale circuit integration, including: Independent Component Analysis (ICA); Brain network topology.
  The above are representative indicators; other relevant brain functional metrics may be included as needed.

SECONDARY OUTCOMES:
Fecal microbiota composition | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session)
  Analysis of the composition and diversity of fecal microbiota (including phylum, genus, and species levels) using high-throughput sequencing of 16S rRNA genes.
Fecal Metabolic Profile | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session)
  Detection of fecal metabolic metabolites (including amino acids, short-chain fatty acids, and bile acids) using liquid chromatography-mass spectrometry (LC-MS) based metabolomics.
Visual Analogue Scale (VAS) for Pain | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assessment of the degree of abdominal pain in participants using a 10-point visual analog scale. Scale Details: Minimum value: 0 points (no pain); Maximum value: 10 points (most severe pain imaginable). Score interpretation: Higher scores indicate more severe abdominal pain.
Short-Form McGill Pain Questionnaire (SF-MPQ) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Evaluates multi-dimensional characteristics of abdominal pain in participants, including pain intensity (assessed via visual analog scale and numerical rating scale) and pain quality (e.g., stabbing, bloating, cramping). Scale Details:
  Minimum value: 0 points; Maximum value: 45 points; Score interpretation: Higher scores indicate more severe and distressing abdominal pain.
Irritable Bowel Syndrome Quality of Life Scale (IBS-QOL) | Baseline (within 1 week before the first TMS session), post-treatment (within 24 hours after the 10th TMS session), 1 month after treatment (±7 days), 3 months after treatment (±7 days)
  Assesses the impact of irritable bowel syndrome on participants' quality of life, covering dimensions such as symptom distress, emotional function, social function, and daily activity limitation. Scale Details: Minimum value: 0 points; Maximum value: 100 points; Score interpretation: Higher scores indicate better quality of life (less impact from IBS symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of Hangzhou Normal University, Hangzhou, Zhejiang, China